CLINICAL TRIAL: NCT03141216
Title: Effects of Mechanical Ventilation on Controlled Volume, Controlled Pressure and Pressure Support in the Immediate Postoperative Period of Cardiac Surgery on Pulmonary Electrical Impedance and Patient-ventilator Asynchrony: a Parallel Clinical Trial
Brief Title: Patient-ventilator Asynchrony in Conventional Ventilation Modes During Short-term Mechanical Ventilation After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Real Hospital Português de Beneficência em Pernambuco (Unknown)
Responsible Party: Principal Investigator, Wagner Souza Leite, Master's Program student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 03021991
Record Dates: First submitted 2017-02-21; First posted 2017-05-05 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: A parallel group study is a simple and commonly used clinical design which compares two treatments. Usually a test therapy is compared with a standard therapy. The allocation of subjects to groups is usually achieved by randomisation. The groups are typically named the treatment group and the control group. Parallel group designs do not require the same number of subjects in each group, although often similar numbers are observed. The design is commonly used in randomised controlled trials. Statistical analysis often boils down to a simple t-test of the between group difference in the outcome, which is usually a mean or a proportion.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCV+PSV (Experimental): volume controlled cycled, assisted-controlled cycled ventilation mode + pressure support ventilation mode. Progression of invasive ventilatory assistance as the patient recovers during post-surgery.
  Interventions: Device: VCV+PSV
- PCV+PSV (Experimental): pressure controlled cycled, assisted-controlled cycled ventilation mode + pressure support ventilation mode. Progression of invasive ventilatory assistance as the patient recovers during post-surgery.
  Interventions: Device: PCV+PSV

INTERVENTIONS:
Device: VCV+PSV — invasive mechanical mechanical modes by volume cycling and by pressure support which the patients will be submitted to before weaning. Post-operative mechanical ventilation average time: 6 hours after ICU admission.
  Other Names: volume controlled ventilation mode; pressure support ventilation mode
  Arms: VCV+PSV
Device: PCV+PSV — invasive mechanical mechanical modes by pressure cycling and by pressure support which the patients will be submitted to before weaning. Post-operative mechanical ventilation average time: 6 hours after ICU admission.
  Other Names: pressure controlled ventilation mode; pressure support mode
  Arms: PCV+PSV

SUMMARY:
This study evaluates the effects of VCV, PCV and PSV ventilatory modes during the immediate postoperative period on the variables resulting from regional and global pulmonary electrical impedance and diaphragmatic mobility, as well as perform ventilator synchrony analysis in PSV mode by mechanical ventilator. Half of the participants will receive VCV followed by PSV for weaning, while the other half will receive PCV followed by PSV for weaning.

DETAILED DESCRIPTION:
In the immediate postoperative period of cardiac surgery, patients are found under mechanical ventilatory support. Commonly, they are ventilated in controlled and assisted-controlled volume (VCV) or pressure (PCV) modes, with weaning at pressure support (PSV).

Systematic reviews indicate that there is no difference between the VCV and PCV ventilatory modes for some clinical outcomes or that the existing evidence is insufficient. The distribution of regional ventilation and diaphragmatic mobility can be measured from the use of electrical impedance tomography (EIT) and diaphragmatic ultrasonography (US) to clarify the physiological changes and / or mechanisms of adaptation of the organism submitted to controlled modes cycled at volume or at pressure and spontaneously flow cycled mode.

Besides EIT and US measures, gasometric, hemodynamic and respiratory data will also be recorded. The statistical analysis will be considered α≤0.05 for a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* IMC 18.5-29.9 kg/m²
* Two thoracic tubes (one mediastinal and one left-sided pleural)
* under mechanical ventilation after surgery
* submitted to intraoperative extracorporeal circulation

Exclusion Criteria:

* Over 2h of cardiopulmonary bypass
* Over 12h of post-operative mechanical ventilation
* Post-operative bleeding above 500 ml in the first hour or above 300 ml in the first two hours
* History of special conditions (neuromuscular and chronic pulmonary disease, thoracic deformity, abdominal distension).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
electrical impedance measures | 5 minutes of recording at each step of mechanical ventilation progression before extubation.
  impedance variation data recorded by a tomograph.

SECONDARY OUTCOMES:
arterial gas blood analysis data | up to 12h, following routine care while patients are mechanically ventilated
  measures of pH, PaCO2 (mmHg), PaO2 (mmHg), PaO2/FiO2
patient-ventilator synchrony | 5 minutes of recording at each step of mechanical ventilation progression before extubation
  events of discomfort between patient and ventilator: ineffective efforts and auto-triggering. Expressed in present or ausent.

CONTACTS AND LOCATIONS:
Overall Officials: WAGNER S LEITE, Principal Investigator — Universidade Federal de Pernambuco; Shirley Lima Campos, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Hospital Real Português de Beneficência em Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
to be shared are: data provided by electrical impedance tomograph, by ultrasound and general clinical one (such as blood pressure, oxygen supplementary concentration, heart rate, respiratory rate, mechanical ventilation duration, surgery duration). These data will be available for sharing after the end of the study and it will be obtained by a copy in a USB flash drive.

REFERENCES:
- See also: Right ventricular function during one-lung ventilation: effects of pressure-controlled and volume-controlled ventilation — http://www.ncbi.nlm.nih.gov/pubmed/24447503
- See also: Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. — https://www.ncbi.nlm.nih.gov/pubmed/9449727
- See also: Tidal ventilation distribution during pressure-controlled ventilation and pressure support ventilation in post-cardiac surgery patients. — https://www.ncbi.nlm.nih.gov/pubmed/25039666
- See also: Monitoring perioperative changes in distribution of pulmonary ventilation by functional electrical impedance tomography. — https://www.ncbi.nlm.nih.gov/pubmed/9689281
- See also: Refining ventilatory treatment for acute lung injury and acute respiratory distress syndrome. — https://www.ncbi.nlm.nih.gov/pubmed/18270359
- See also: Bedside waveforms interpretation as a tool to identify patient-ventilator asynchronies. — https://www.ncbi.nlm.nih.gov/pubmed/16283171
- See also: Volume-controlled versus pressure-controlled ventilation-volume guaranteed mode during one-lung ventilation — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4216788/
- See also: Ultrasonographic diagnostic criterion for severe diaphragmatic dysfunction after cardiac surgery. — https://www.ncbi.nlm.nih.gov/pubmed/18753469
- Available data/document: Study Protocol — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Search for "buscar pesquisas aprovadas" and fill the the blanks with research title and investigator's full name